CLINICAL TRIAL: NCT00468039
Title: A Multicenter, Open-label Sub-study to LMF237A2302 to Assess the Effect of 24 Weeks Treatment With Initial Combination of Vildagliptin 100mg qd Plus Metformin 1000mg Bid in Drug Naive Patients With Type 2 Diabetes With Very Poor Glycemic Control
Brief Title: A Sub-study to LMF237A2302 to Assess the Effect of 24 Weeks Treatment With Initial Combination of Vildagliptin Plus Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLMF237A2302S1
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: metformin; vildagliptin; initial combination
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin

ARMS (1):
- vildagliptin + metformin (Experimental)
  Interventions: Drug: vildagliptin + metformin

INTERVENTIONS:
Drug: vildagliptin + metformin

SUMMARY:
This study will evaluate the effects of treatment with vildagliptin and metformin as initial combination in newly diagnosed patients with type 2 diabetes who have very high levels of HbA1c and/or fasting plasma glucose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (non-fertile or of childbearing potential using a medically approved birth control method) patients with type 2 diabetes
* Diagnosis of type 2 diabetes for at least 4 weeks prior to study entry
* Body mass index 22-40 kg/meter squared
* HbA1c > 11% and/or FPG >270 mg/dL

Exclusion Criteria:

* Pregnant or lactating female
* History of type 1 diabetes
* Evidence of significant diabetic complications
* Treatment with insulin or any other oral antidiabetic agent

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-03-06 (Actual); Primary Completion 2008-06-06 (Actual); Study Completion 2008-06-06 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin (HbA1c)at Baseline and week 24 | 24 weeks

SECONDARY OUTCOMES:
HbA1c at Baseline and week 12 | 12 weeks
Fasting plasma glucose test (FPG) at Baseline and week 24 | 24 weeks
Weight at baseline and week 24 | 24 weeks
Responder rates assessed by HbA1c absolute reduction from baseline to endpoint greater than or equal to 0.7% after 24 weeks | 24 weeks
Safety assessed by monitoring and recording all adverse events, serious adverse events. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Diabetes and Glandular Disease Research Associates, San Antonio, Texas, United States

REFERENCES:
- [Result] Bosi E, Dotta F, Jia Y, Goodman M. Vildagliptin plus metformin combination therapy provides superior glycaemic control to individual monotherapy in treatment-naive patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2009 May;11(5):506-15. doi: 10.1111/j.1463-1326.2009.01040.x. Epub 2009 Mar 23. PMID 19320662
- See also: Results for CLMF237A2302S1 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2651